CLINICAL TRIAL: NCT01298076
Title: A Multicentre Randomised Clinical Trial of Intravitreal Bevacizumab (Avastin®) Versus Intravitreal Dexamethasone (Ozurdex™) for Persistent Diabetic Macular Oedema
Brief Title: Intravitreal Bevacizumab (Avastin®) Versus Intravitreal Dexamethasone (Ozurdex™) for Persistent Diabetic Macular Oedema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Mark Gillies, Professor, University of Sydney
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHMRC project 632667; 2009-01024 (Other Grant/Funding Number: NHMRC-PROJECT GRANT ACCEPTANCE-RIMS Project ID)
Record Dates: First submitted 2010-08-31; First posted 2011-02-17 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Diabetic Retinopathy; Macular Edema
Keywords: Diabetes; Retinopathy; Macular oedema; Laser; Photocoagulation; Fovea; Steroid; Bevacizumab; Intravitreal
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema; Diabetes Mellitus; Retinal Diseases | interventions — Bevacizumab; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AVASTIN (Active Comparator): intravitreal bevacizumab
  Interventions: Drug: bevacizumab
- OZURDEX (Active Comparator): intravitreal dexamethasone
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: bevacizumab — Anti-VEGF drug for intravitreal injection
  Arms: AVASTIN
Drug: dexamethasone — Slow-release steroid formulation for intravitreal injection
  Arms: OZURDEX

SUMMARY:
The specific aims of the study are to test the following hypotheses:

* That there is a difference in change in visual acuity resulting from treatment with intravitreal bevacizumab compared with dexamethasone implant in eyes with advanced macular oedema
* That there is a difference in degree of resolution of macular oedema resulting from treatment with intravitreal bevacizumab compared with dexamethasone implant in eyes with advanced macular oedema
* That both intravitreal bevacizumab and dexamethasone implants have a manageable and acceptable safety profile in eyes with diabetic macular oedema

DETAILED DESCRIPTION:
Diabetic retinopathy is a common cause of severe loss of vision and the most common cause of blindness in individuals between the ages of 20 and 65 years in developed countries. Swelling of the central retina, or "macular oedema", is the commonest cause of visual loss in diabetic retinopathy.

Diabetic macular oedema (DMO) is treated with laser photocoagulation of areas of leak in the macula according to established guidelines which take into account the extent of the leak and its proximity to the centre of the macula, the "fovea". This treatment does not always work, however, and is inherently destructive.

New drugs have become available which appear to reduce the risk of loss of vision in eyes with advanced diabetic macular oedema for which further laser treatment is unlikely to be beneficial. Intravitreal injection of slow-release steroid formulations such as Ozurdex™, a slow release formulation of dexamethasone, has been proposed as a new modality to treat clinically significant DMO. We have recently conducted randomised clinical trials which have demonstrated that treatment with intravitreal triamcinolone (IVTA) leads to reduction of DMO and improved vision in these eyes. Another class of drugs, inhibitors of Vascular Endothelial Growth Factor (VEGF) such as bevacizumab (Avastin®), also appear efficacious.

While both drugs appear to reduce macular oedema and improve vision in the short term, they may have differences which could guide how they are best used. Around 1/3 of eyes that receive dexamethasone may develop elevated intraocular pressure and cataract, both of which are manageable but may complicate the picture. Anti-VEGF drugs do not have these local adverse events, however they must be given more frequently (4-6 weekly vs 4-6 monthly for Ozurdex™) and it is suspected they may have a neurotoxic effect on the retina. Some authorities suspect that anti-VEGF treatment may be associated with a small increased risk of having a stroke or heart attack during treatment, even when they are injected into the eye. This has not been proven with a related drug, ranibizumab, but it is still possible that it may occur with bevacizumab.

This will be a, 2 year, phase II, prospective, multicentre, randomised, single-masked clinical trial of sustained release intravitreal dexamethasone (Ozurdex™) versus intravitreal injections of bevacizumab (Avastin®) for diabetic foveal oedema that persists or recurs despite previous laser treatment, or for which the investigator believes laser treatment is unlikely to be helpful.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Diagnosis of diabetes mellitus types 1 or 2
* Diabetic macular oedema affecting the fovea in one or both eyes (phakic or pseudophakic) for which laser treatment is unlikely to be helpful in the opinion of the centre chief investigator
* Best corrected visual acuity of 17-72 letters (6/12 -6/120)
* Retinal thickness > 250 micron in central 1mm subfield on Stratus (time domain) OCT and 300 on Spectral domain OCT
* Previous macular laser treatment, or the investigator believes laser treatment is unlikely to be helpful
* Intraocular pressure <22mmHg
* Women of childbearing potential must have a negative urine pregnancy test at the screening visit and prior to treatment. A woman is considered of childbearing potential unless she is postmenopausal and without menses for 12 months or is surgically sterilised
* Written informed consent has been obtained.

Exclusion Criteria:

* Known allergy to Ozurdex, Avastin or agents used in the study
* Women who are pregnant, nursing, or planning a pregnancy, or who are of childbearing potential and not using reliable means of contraception
* Glaucoma which is uncontrolled or is controlled but with more than one medication or with only one medication and with glaucomatous field defects
* Loss of vision due to other causes (e.g. age related macular degeneration, myopic macular degeneration, retinal vein occlusion)
* Macular oedema due to other causes
* An ocular condition that would prevent visual acuity improvement despite resolution of oedema (such as foveal atrophy or substantial premacular fibrosis)
* Treatment with IVTA within the last 6 months or peribulbar TA within the last 3 months or bevacizumab within the last 2 months.
* Cataract surgery within the last 6 months
* Retinal laser treatment within the last 3 months
* History of herpes virus infection in study eye
* Media opacity including cataract that already precludes adequate macular photography and laser treatment, or cataract that is likely to require surgery within 2 years
* Known allergies to dexamethasone or bevacizumab
* Patient is already receiving systemic steroid treatment > 5mg prednisolone daily or equivalent)
* Intercurrent severe disease such as septicemia, any condition which would affect follow-up or photographic documentation (e.g. geographical, psycho-social)
* History of chronic renal failure requiring dialysis or renal transplant
* Blood pressure >180/110
* Patient has a condition or is in a situation that in the investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Visual acuity gain | 2 years
  The comparison of the proportion of eyes gaining 10 letters of visual acuity between the bevacizumab (Avastin®) and dexamethasone (Ozurdex™) implant arms after 104 weeks.

SECONDARY OUTCOMES:
Visual acuity change | 2 years
  Change in visual acuity compared with the pre-injection level
OCT change | 2 years
  Change in retinal thickness demonstrated on optical coherence tomography(OCT)
Laser requirement | 2 years
  Number of laser treatments required for the treatment of macular oedema
Patient satisfaction | 2 years
  Patient satisfaction with treatment
Safety | 2 years
  * Mean change in maximum diameter of foveal avascular zone
  * Incidence and severity of ocular adverse events
  * Incidence and severity of non ocular adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Gillies, Professor, Principal Investigator — University of Sydney
Locations (4):
- Australia (4):
  - Save Sight Institute, Sydney, New South Wales
  - South West Retina, Sydney, New South Wales
  - Centre for Eye Research Australia, Melbourne, Victoria
  - Lions Eye Institute, Perth, Western Australia

REFERENCES:
- [Derived] Rittiphairoj T, Mir TA, Li T, Virgili G. Intravitreal steroids for macular edema in diabetes. Cochrane Database Syst Rev. 2020 Nov 17;11(11):CD005656. doi: 10.1002/14651858.CD005656.pub3. PMID 33206392
- [Derived] Mehta H, Fraser-Bell S, Nguyen V, Lim LL, Gillies MC. The Interval between Treatments of Bevacizumab and Dexamethasone Implants for Diabetic Macular Edema Increased over Time in the BEVORDEX Trial. Ophthalmol Retina. 2018 Mar;2(3):231-234. doi: 10.1016/j.oret.2017.06.010. Epub 2017 Aug 23. PMID 31047591
- [Derived] Mehta H, Fraser-Bell S, Nguyen V, Lim LL, Gillies MC. Short-term vision gains at 12 weeks correlate with long-term vision gains at 2 years: results from the BEVORDEX randomised clinical trial of bevacizumab versus dexamethasone implants for diabetic macular oedema. Br J Ophthalmol. 2018 Apr;102(4):479-482. doi: 10.1136/bjophthalmol-2017-310737. Epub 2017 Aug 4. PMID 28779007
- [Derived] Wickremasinghe SS, Fraser-Bell S, Alessandrello E, Mehta H, Gillies MC, Lim LL. Retinal vascular calibre changes after intravitreal bevacizumab or dexamethasone implant treatment for diabetic macular oedema. Br J Ophthalmol. 2017 Oct;101(10):1329-1333. doi: 10.1136/bjophthalmol-2016-309882. Epub 2017 Feb 22. PMID 28228411
- [Derived] Aroney C, Fraser-Bell S, Lamoureux EL, Gillies MC, Lim LL, Fenwick EK. Vision-Related Quality of Life Outcomes in the BEVORDEX Study: A Clinical Trial Comparing Ozurdex Sustained Release Dexamethasone Intravitreal Implant and Bevacizumab Treatment for Diabetic Macular Edema. Invest Ophthalmol Vis Sci. 2016 Oct 1;57(13):5541-5546. doi: 10.1167/iovs.16-19729. PMID 27768792
- [Derived] Mehta H, Fraser-Bell S, Yeung A, Campain A, Lim LL, Quin GJ, McAllister IL, Keane PA, Gillies MC. Efficacy of dexamethasone versus bevacizumab on regression of hard exudates in diabetic maculopathy: data from the BEVORDEX randomised clinical trial. Br J Ophthalmol. 2016 Jul;100(7):1000-1004. doi: 10.1136/bjophthalmol-2015-307797. Epub 2015 Nov 4. PMID 26537156
- [Derived] Gillies MC, Lim LL, Campain A, Quin GJ, Salem W, Li J, Goodwin S, Aroney C, McAllister IL, Fraser-Bell S. A randomized clinical trial of intravitreal bevacizumab versus intravitreal dexamethasone for diabetic macular edema: the BEVORDEX study. Ophthalmology. 2014 Dec;121(12):2473-81. doi: 10.1016/j.ophtha.2014.07.002. Epub 2014 Aug 22. PMID 25155371